CLINICAL TRIAL: NCT05678127
Title: Skin Biopsy as Diagnostic Tool in Anterior Cutaneous Nerve Entrapment Syndrome (ACNES): A Pilot Study
Brief Title: A Pilot Study to Explore the Use of Skin Biopsy as Diagnostic Tool in Anterior Cutaneous Nerve Entrapment Syndrome (ACNES)
Acronym: Biopsy-ACNES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, dr. RMH Roumen, surgeon, Head of surgery, Principal Investigator, Maxima Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL81661.015.22
Record Dates: First submitted 2022-12-29; First posted 2023-01-10 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Anterior Cutaneous Nerve Entrapment Syndrome; Nerve Entrapment Syndrome; Chronic Pain Syndrome; Diagnosis
Keywords: Diagnostic test for ACNES; Intraepidermal nerve fibre density (IENFD)
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Disease

STUDY DESIGN:
Intervention Model Description: Skin biopsies will be performed on patients with an unilateral ACNES. Biopsies will be taken at the triggerpoint (affected side) and contralateral, non-affected side of the abdominal wall.
  Affected vs non-affected will be compared. The non-affected side serves as control.
Masking Description: The pathologists who will measure the nerve fibre density are blinded; they will not know if the biopsy is from the affected or non-affected side.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with unilateral ACNES (Experimental)
  Interventions: Procedure: Skin biopsy

INTERVENTIONS:
Procedure: Skin biopsy — Two 3mm skin biopsies from the abdominal wall will be taken. One at the triggerpoint of the pain, the second one at the contralateral, non-affected side of the abdominal wall.
  Lidocaine will be used for local anaesthesia of the skin, before the biopsies will be taken.

SUMMARY:
ACNES is a neuropathic pain condition of the abdominal wall. It is a clinical diagnosis based on patient's history and physical examination. No diagnostic test is available to confirm the diagnosis.

This pilot study will determine if skin biopsies can be used as diagnostic test. Two 3mm biopsies will be taken and used to count the small nerve fibres in the skin. The number of small nerve fibres of the painful skin will be compared to non-painful skin. Skin biopsy and small fibre nerve count is already used as diagnostic test in patients with small-fibre neuropathy.

The investigators hypothesize that patients with ACNES will have a reduced number of small nerve fibres in the affected skin, compared to the non-affected skin.

ELIGIBILITY:
Inclusion Criteria:

* Duration of pain >3 months
* Newly diagnosed unilateral ACNES
* Fully completed intake questionnaire
* Obtained written informed consent

Exclusion Criteria:

* Inability to understand Dutch language
* Bilateral ACNES
* Previously administered injections with corticosteroids at trigger point (injection with a local anaesthetic is allowed)
* Previous Pulsed Radiofrequency (PRF)-treatment at trigger point
* History of open abdominal surgery
* History of neurectomy
* Known neuromuscular or neurodegenerative disease
* Antiplatelet or anticoagulants use or known coagulation disorders
* Disorder known to cause a reduced IENFD;

  * Diabetes
  * Hypothyroidism
  * Renal failure
  * Vitamin B12 deficiency
  * Monoclonal gammopathy
  * Alcohol abuse (>5 IU a day)
  * Malignancies
  * Medication that cause neuropathy (for example chemotherapy)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Intraepidermal Nerve Fibre density (IENFD) | Both biopsies will be taken at the same time, as their difference will be studied. The biopsies will be taken at the second outpatient visit, 2 or 3 weeks after the first visit, just after the second triggger point injection (standard of care).
  Difference in IENFD (measured in IENF/mm) from both affected and non-affected side of the abdominal wall.

SECONDARY OUTCOMES:
Pain score | Assessed at first outpatient visit, used as baseline data.
  Average pain score, assessed using the Numeric Rating Scale (NRS) 0-10 before start of treatment. 0 no pain, 10 worst possible pain.
Duration of pain | Assessed at first outpatient visit, used as baseline data.
  Duration of pain in months before diagnosis
Treatment response | Treatment response will be assessed 2 to 6 weeks after each treatment (trigger point injections, PRF and neurectomy), as standard of care.
  Patients will receive standard of care treatment for ACNES. Treatment is unsuccessful if <50% pain reduction or when patients are not satisfied with their pain relief and want additional treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rudi Roumen, MD, PhD, Principal Investigator — Maxima Medical Center
Locations (1):
- Maxima Medical Center, Veldhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided